CLINICAL TRIAL: NCT00826319
Title: CanPREDDICT: Canadian Study of Prediction of Risk and Evolution to Dialysis, Death and Interim Cardiovascular Events Over Time
Brief Title: Canadian Study of Prediction of Risk and Evolution to Dialysis, Death and Interim Cardiovascular Events Over Time
Acronym: CanPREDDICT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: H07-02457
Record Dates: First submitted 2009-01-20; First posted 2009-01-22 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-11

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic Kidney Disease; Renal Insufficiency; Biomarkers; Observational
MeSH Terms: conditions — Renal Insufficiency, Chronic; Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum,Plasma,Urine, DNA and RNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Bioimpedance sub-study cohort: Funded by a grant from Kidney Foundation of Canada, Dr. Catherine Clase initiated a bioimpedance sub-study across 7 centres and recruited n=416 within the CANPREDDICT population. The study uses bioimpedance measurements to assess volume status to determine the multivariable relationship between baseline volume overload and subsequent cardiovascular events. Subjects are followed at 6 months intervals for 2 years.
- Ethnic enrichment cohort: Additional recruitment initiated and funded by the Principal Investigator, Adeera Levin for enriching the ethnic representation within the Canadian cohort on South Asian and Oriental Asian was completed from Sept 2012 to June 2013, n=53.
- Original CanPreddict cohort: The original CanPreddict cohort was recruited from Jun 2008 - Oct 2009 has 2544 CKD patients across Canada.

SUMMARY:
This study will follow 2500 prevalent Chronic Kidney Disease (CKD) patients with Glomerular Filtration Rate (GFR) from 15-45 ml/min for 30 months with serial measurements every 6 months and subsequent annual chart review up to 60 months. This observational study will analyze the demographics, clinical status, medications and blood and urine samples of these patients and study the conventional biochemical, hormonal and metabolic parameters assessing which underlying biomarkers reflect the processes involved with disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients currently seen by a nephrologist, or referred for evaluation of CKD
* GFR between 15-45 ml/min
* Adults 19 years (depending on age of consent in province) or older
* At pediatric sites study participants will be eligible to participate at age 15 or older

Exclusion Criteria:

* Organ transplant recipient
* Life expectancy less than 12 months
* Acute Vasculitis
* Bioimpedance sub-study exclusion criteria:
* Amputation (readings are inaccurate)
* Any battery operated or electronic implanted device (such as pacemaker or implanted defibrillator - potential electrical hazard)
* Pregnant women

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Nephrology Clinics across Canada
Sampling Method: Non-Probability Sample
Enrollment: 2602 (Actual)
Dates: Start 2008-06; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Renal Replacement Therapy | 6 monthly for 3 years, annually up to 5 years
  Renal Replacement Therapy is defined as dialysis start or transplantation.
Cardiovascular events | 6 monthly for 3 years, annually up to 5 years
  Cardiovascular events are defined as myocardial infarction, ischemic and hemorrhagic stroke, coronary revascularization, congestive heart failure, peripheral bypass and gangrenes, adjudicated by a nephrologist, cardiologist and neurologist.
Death | 6 monthly for 3 years, annually up to 5 years
  Deaths are reported with source documentation and adjudicated for ischemic or congestive cardiovascular death, other cardiovascular death, non-cardiovascular death and unknown cause of death.

CONTACTS AND LOCATIONS:
Overall Officials: Adeera Levin, Principal Investigator — University of British Columbia
Locations (25):
- Canada (25):
  - Foothills Hospital, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Penticton Regional Hospital, Penticton, British Columbia
  - BC Children's Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Eastern Regional Health Authority, Health Sciences Centre, St. John's, Newfoundland and Labrador
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Cape Breton District Health Authority, Sydney, Nova Scotia
  - St Joseph's Hospital, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - London Health Science Centre- University Campus, London, Ontario
  - London Health Science Centre- Victoria Campus, London, Ontario
  - York Central, Oak Ridges, Ontario
  - University of Ottawa, Ottawa, Ontario
  - Timmins & District Hospital, Timmins, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Sunnybrook Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Charles Le Moyne Hospital, Greenfield Park, Quebec
  - Hôpital du Sacré-Coeur, Montreal, Quebec
  - Maisonneuve-Rosemont Hopital, Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec
  - CHUQ: L'Hôtel-Dieu de Québec, Québec, Quebec

REFERENCES:
- [Result] Levin A, Rigatto C, Brendan B, Madore F, Muirhead N, Holmes D, Clase CM, Tang M, Djurdjev O; CanPREDDICT investigators. Cohort profile: Canadian study of prediction of death, dialysis and interim cardiovascular events (CanPREDDICT). BMC Nephrol. 2013 Jun 11;14:121. doi: 10.1186/1471-2369-14-121. PMID 23758910
- [Result] Levin A, Rigatto C, Barrett B, Madore F, Muirhead N, Holmes D, Clase C, Tang M, Djurdjev O. (2012). Canadian study of prediciont of death, dialysis and interim cardiovascular events: CanPREDDICT: Biomarkers improve prediction of one year outcomes in chronic kidney disease cohort. Clinical studies in CKD. Nephrology Dialysis Transplantation, 27(suppl 2), ii63-ii65.
- [Result] Levin A, Rigatto C, Barrett B, Madore F, Muirhead N, Holmes D, Clase CM, Tang M, Djurdjev O; CanPREDDICT Investigators. Biomarkers of inflammation, fibrosis, cardiac stretch and injury predict death but not renal replacement therapy at 1 year in a Canadian chronic kidney disease cohort. Nephrol Dial Transplant. 2014 May;29(5):1037-47. doi: 10.1093/ndt/gft479. Epub 2013 Dec 26. PMID 24371297